CLINICAL TRIAL: NCT01020084
Title: Effect of Hyposalivation on Mastication and Speech
Brief Title: Salivary Flow Rate and Oral Function
Acronym: SOF
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Renata Cunha Matheus Rodrigues Garcia, Piracicaba Dental School, State University of Campinas
Other Study IDs: monegfg09
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Food Comminution; Jaw Movements
Keywords: Saliva; Mastication; Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Subjects with normal salivary flow rate
- Hyposalivation: Subjects presenting low salivary flow rate as a side effect of systemic isotretinoin therapy.

SUMMARY:
The purpose of this study was to investigate if salivary flow rate is important to maintain adequate oral functions.

DETAILED DESCRIPTION:
Hyposalivation may damage oral functions. Therefore, the aim of this study was to evaluate whether patients under hyposalivation present damaged mastication and speech. Forty subjects composed 2 groups: Control (C) and hyposalivation (H). Masticatory performance (MP) was carried out using artificial material and a 10-sieve method. Mandibular movements during speech were obtained using a 3D jaw-tracking device. Neither mastication nor speech have been impaired by low salivary flow rate.

ELIGIBILITY:
Inclusion Criteria:

* Fully dentate
* Good general and oral health

Exclusion Criteria:

* Signs or symptoms of temporomandibular disorders
* Parafunctions
* Malocclusion
* History of communication deficits or prior speech-language treatment

Ages: 16 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Forty subjects were selected (20 male and 20 female) among people seeking for dental treatment, students and staff of Piracicaba Dental School.Saliva collection was performed for all subjects, and indivuduals with normal salivary flow rate composed the control group. Hyposalivation group group, otherwise, was composed by subjects taking 0.5-0.7 mg/kg/day for at least one month prescribed by a dermatologist.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-08; Primary Completion 2006-08 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renata CM Rodrigues Garcia, PhD, Study Chair — Piracicaba Dental School; Alrair A Del Bel Cury, PhD, Study Director — Piracicaba Dental School; Simone G Farias Gomes, MS, Principal Investigator — Piracicaba Dental School
Locations (1):
- Piracicaba Dental School, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Background] Saliva: its role in health and disease. Working Group 10 of the Commission on Oral Health, Research and Epidemiology (CORE). Int Dent J. 1992 Aug;42(4 Suppl 2):287-304. No abstract available. PMID 1399047
- [Background] Bianchini EM, de Andrade CR. A model of mandibular movements during speech: normative pilot study for the Brazilian Portuguese language. Cranio. 2006 Jul;24(3):197-206. doi: 10.1179/crn.2006.032. PMID 16933461
- [Result] Liedberg B, Owall B. Masticatory ability in experimentally induced xerostomia. Dysphagia. 1991;6(4):211-3. doi: 10.1007/BF02493529. PMID 1778098
- [Result] Ishijima T, Koshino H, Hirai T, Takasaki H. The relationship between salivary secretion rate and masticatory efficiency. J Oral Rehabil. 2004 Jan;31(1):3-6. doi: 10.1111/j.1365-2842.2004.01033.x. PMID 15125589